CLINICAL TRIAL: NCT03328793
Title: Musicians United for Seniors to Improve Care (MUSIC) Study - Open Randomized Controlled Clinical Trial Examining the Effect of Live Music Sessions on Health Condition of Geriatric Inpatients
Brief Title: Musicians United for Seniors to Improve Care (MUSIC) Study
Acronym: MUSIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Shek Fung, Principal Investigator, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SMHC 14-31B
Record Dates: First submitted 2017-10-13; First posted 2017-11-01 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Music; Gait; Emotions; Communication
Keywords: music; gait; emotions; communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research assistant who will be doing the Visual Analog Mood Scale (VAMS) with the patients pre and post intervention will be blinded in regards to the group attribution of the patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Intervention (Intervention Group) (Experimental): The patients will assist to a live music session of 30 minutes which will be given by musicians (volunteers) and will undergo:
  * mood assessment
  * emotion assessment
  * mobility assessment
  * communication assessment
  Interventions: Behavioral: Mood Assessment; Behavioral: Emotion Assessment; Behavioral: Communication Assessment; Other: Mobility assessment; Other: Music Intervention
- Documentary watching (Control Group) (Active Comparator): The patients will watch a documentary for 30 minutes in the presence of a volunteer and will undergo:
  * mood assessment
  * emotion assessment
  * mobility assessment
  * communication assessment
  Interventions: Behavioral: Mood Assessment; Behavioral: Emotion Assessment; Behavioral: Communication Assessment; Other: Mobility assessment; Other: Documentary watching

INTERVENTIONS:
Behavioral: Mood Assessment — Prior to and after the session, the patients will be asked to fill a VAMS (Visual Analog Mood Scale).
Behavioral: Emotion Assessment — During the sessions, the patients will be videotaped and the videotapes will be reviewed by 2 independent research assistants. With the use of the Observed Emotional Rating Scale (OERS), the research assistants will be able to assess the patients's emotions at the beginning and at the end of the session (they will analyse the first 10 and the last 10 minutes of the sessions).
Behavioral: Communication Assessment — During the sessions, the patients will be videotaped and the videotapes will be reviewed by 2 independent research assistants. With the use of the CODEM Scale, the research assistants will be able to assess the patients's emotions at the beginning and at the end of the session (they will analyse the first 10 and the last 10 minutes of the sessions).
Other: Mobility assessment — If deemed to be safe, the patients will undergo a gait speed assessment as well as a TUG (timed-up-and-go) prior to and after the sessions
Other: Music Intervention — The participants will listen to a 30 minute live music sessions which will be given by musicians (who is a volunteer)
  Arms: Music Intervention (Intervention Group)
Other: Documentary watching — The patients will watch a documentary for 30 minutes in the presence of a volunteer
  Arms: Documentary watching (Control Group)

SUMMARY:
Music has a potential role in health care. In the geriatric population, music presents a non-pharmacological intervention which is easy to implement. Also, music has a potential role in order to improve patient's mobility. For example, it was also shown that the rhythmic component of music combined with physical exercise can improve gait variability which has been identified as a marker of gait instability and a fall predictor. This effect was previously shown in older community dwellers as a music-based intervention significantly improved gait and balance stability.

Considering that music was shown to have a positive impact on communication, emotions and depressive symptoms this intervention has the potential to make our patients more conscious of their environment, leading to an improved mobility.

Thus, the investigators hypothesize that patients who attend live music sessions (compared to controls) will demonstrate an improvement in their mobility measures. This effect could potentially be explained by the rhythmic effect of music and by the fact that live music sessions lead to an improved mood, communication, emotions, and an improved mobility.

* The primary objective of this study will be to determine if participation to live music sessions will be associated with an improvement in mobility which will be measured using the Times Up and Go (TUG) and gait speed when compared to a control group.
* The second objective of this study will be to determine if patients participating in live music sessions compared to a control group demonstrate an increase/improvement at the end of their music session in their mood (the Visual Analog Mood Scale (VAMS) will be used), in their positive emotions (the Observed Emotion Rating Scale (OERS) will be used) and communication behaviour (the CODEM (tool to assess communication behavior in dementia) instrument will be used).
* The third objective of this study will be to perform a "feasibility study". By measuring the variation in the different scales which will be used (see the third objective), the investigators will be able to determine how many participants will be necessary for an eventual larger scale study.

This will be a prospective open-label randomized control trial. The patients will be randomly assigned to a musical intervention or to a television intervention (control group). The patients will only attend one session in the context of this research project. Pre and post measures will be done.

DETAILED DESCRIPTION:
Music has a potential role in health care. In patients with major neurocognitive impairment (previously called dementia), several studies have demonstrated that musical intervention can improve cognition, in particular spatial and temporal orientation, episodic memory and working memory. It was also shown that music may improve quality of life and reduce depressive symptoms, and there is growing evidence for the use of music to treat pain and anxiety.

When specifically looking at the geriatric population, music listening presents a non-pharmacological intervention which is easy to implement in inpatients with functional decline. It was shown to improve mood in both cognitively impaired and intact patients.

Music has a potential role in order to improve patient's mobility. For example, it was also shown that the rhythmic component of music combined with physical exercise can improve gait variability which has been identified as a marker of gait instability and a fall predictor. This effect was previously shown in older community dwellers as a music-based intervention significantly improved gait and balance stability.

Also, considering that music was shown to have a positive impact on communication, emotions and depressive symptoms, this intervention therefore has the potential to make our patients more conscious of their environment, leading to an improved mobility.

Thus, the investigators hypothesize that patients who attend live music sessions (compared to controls) will demonstrate an improvement in their mobility measures. This effect could potentially be explained by the rhythmic effect of music and by the fact that live music sessions lead to an improved mood, communication, emotions, and an improved mobility.

* The primary objective of this study will be to determine if participation to live music sessions will be associated with an improvement in mobility which will be measured using the Times Up and Go (TUG) and gait speed when compared to a control group.
* The second objective of this study will be to determine if patients participating in live music sessions compared to a control group demonstrate an increase/improvement at the end of their music session in their mood (the Visual Analog Mood Scale (VAMS) will be used), in their positive emotions (the Observed Emotion Rating Scale (OERS) will be used) and communication behaviour (the CODEM instrument will be used).
* The third objective of this study will be to perform a "feasibility study". By measuring the variation in the different scales which will be used (see the third objective), the investigators will be able to determine how many participants will be necessary for an eventual larger scale study.

This will be a prospective open-label randomized control trial. The patients will be randomly assigned to a musical intervention or to a television intervention (control group). The patients will only attend one session in the context of this research project. Pre and post measures will be done.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Geriatric Assessment Unit of St. Mary's Hospital.
* Patients interested in participating in this research (recreational) study

Exclusion Criteria:

* Patients who are medically unstable to attend the music or television-watching sessions will be excluded from the study.
* Also, if patients are deemed to be unsafe by the medical team to undergo a TUG or a gait speed assessment, those measures will not be collected. Those patients would therefore only fill a pre- and post VAMS and attend the musical or television session.
* Finally, the investigators will only consider the first participation to a session in our analysis. In other words, patients who have already participated to a music session prior to the initiation of this study will be excluded (will not be recruited into the study).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Timed up and Go (measured in seconds) compared to after completion of the session. | At baseline (T0), and within 5 minutes of completion of the intervention session (T1)
  Measure of mobility, uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. Has excellent interrater (intraclass correlation coefficient [ICC] = .99) and intrarater reliability (ICC = .99)
Change from baseline Gait speed (measured in seconds) compared to after completion of the session. | At baseline (T0), and within 5 minutes of completion of the intervention session (T1)
  Measure of mobility, measures time that a person takes to walk 3 meters at their comfortable pace in a quiet, well-lit corridor wearing their own footwear. In order to avoid acceleration and deceleration effects, participants will start walking one meter before the "start line" and will walk one meter beyond the "finish line".

SECONDARY OUTCOMES:
Change from baseline Visual Analog Mood Scale compared to after completion of the session. | At baseline (T0), and within 5 minutes of completion of the intervention session (T1)
  Evaluation of 8 moods (happy, afraid, confused, sad, angry, energetic, tired and tense) with the use of schematic faces connected by a 100-mm vertical line. The top picture depicts a neutral mood face, while each of the eight scales are depicted below. The patients are asked to draw a line across the 100-mm vertical line to represent their current mood state.
Change in the Observed Emotional Rating Scale at the beginning of the session compared to the end of the session. | Start of intervention session and end of intervention session (i.e the first 10 minutes and last 10 minutes of videotaped sessions)
  Consists of an observational tool including 2 positive emotions (pleasure and general alertness) and three negative emotions (anger, anxiety/fear, and sadness). The duration of each affect is measured over a ten-minute period and is graded from 1 to 5 (1 =never, 2 < 16 seconds, 3 = 16-59 seconds, 4 = 1-4 minutes, and 5 = >5 minutes).
  Will be used to code the first 10 minutes and last 10 minutes of videotaped sessions.
Change in Communication Skills at the beginning of the session compared to the end of the session. | Start of intervention session and end of intervention session (i.e the first 10 minutes and last 10 minutes of videotaped sessions)
  The CODEM (tool to assess communication behavior in dementia) scales will be used. This scale requires a 10-minute observation-period of the participant and uses a scale from 0 to 5 to quantify the communication skills of the participants from 0 to 5 (0 = behavior is not shown during the interaction, 1 = behavior is rarely seen (1-24% during the interaction), 2 = behavior is shown in less than half (25-49%) of the interaction, 3 = behavior is shown in more than half (51-75%) of the interaction, 4 = behavior is shown in almost all (76-99%) interaction situations, and 5 = behavior is always shown (100%) during the interaction). It consists of 15 different items (8 verbal and 7 non-verbal items). For example, eye contact is a non-verbal item.
  Will be used to code the first 10 minutes and last 10 minutes of videotaped sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Mary's Hospital Center, Montreal, Quebec, Canada